CLINICAL TRIAL: NCT04785248
Title: A Prospective Clinical Observation of Ventriculo-Peritoneal Shunt in Patients With Normal or Low Hydrocephalus and A Multi-Center Randomized Controlled Study on Application of "Three-step Disinfection" in Reducing the Incidence of Post-operative Infection
Brief Title: Clinical Observation of V-P Shunt and Application of "Three-step Disinfection" to Reduce Post-operative Infection Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baiyun Liu (Other)
Responsible Party: Sponsor-Investigator, Baiyun Liu, Professor, Chief Physician, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BTHospital HX-A-035(2020); BTHospital KY2021-016-03 (Other: IRB of Beijing Tiantan Hospital)
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Hydrocephalus; Ventriculoperitoneal Shunt
Keywords: Ventriculoperitoneal Shunt; Surgical Wound Infection; Disinfection
MeSH Terms: conditions — Hydrocephalus; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled group (No Intervention): the routine preoperative disinfection method
- Three-step disinfection (Experimental): new developed method of preoperative disinfection
  Interventions: Procedure: Three-step disinfection

INTERVENTIONS:
Procedure: Three-step disinfection — Three step disinfection method can be divide in three part. The first step of disinfection: scalp dandruff removal + disinfection The second step of disinfection: whole head Use 2% iodine tincture to smear the whole head skin, the assistant helps to lift the head to expose the surgical field, from both eyebrows to the occipital hairline, from both sides to the neck, after the iodine tincture dry out, use 75% alcohol to deionize. Then placing more than 4 layers of operation towel under the head.
  The third step of disinfection: neck chest abdomen disinfection.
  Arms: Three-step disinfection

SUMMARY:
A randomized, single blind, parallel controlled, multicenter clinical study was performed in which patients who had undergone a cerebrospinal fluid to peritoneal shunt that met the criteria were divided into two groups (test and control) in a 1:1 ratio, with the test group applied disinfection by the "three-step sterilization method" and completed the procedure, and the control group underwent the same surgical procedure according to the routine aseptic disinfection procedure, relevant literatures were reviewed and the previous ones in our hospital were summarized, it is intended to conduct a one-year clinical observation of the two groups, to compare the perioperative and long-term infection incidence of the two groups and evaluate them comprehensively, to evaluate whether the "three-step sterilization method" disinfected patients have reduced perioperative and long term infection risk after surgery compared with previous surgery with routine disinfection procedure, and to evaluate their effectiveness.

DETAILED DESCRIPTION:
Data Collection:

Preoperative symptoms and signs, medical records, imaging data, preoperative functional scores (Glasgow score, ADL score, jnphgsr score) were collected.

Data Security Monitoring:

1. Follow-up after surgery according to the study scheme, and comprehensive collection of safety data, for key patient researchers should focus on, in order to comprehensively and early detection of all kinds of adverse events.
2. All adverse events are well documented, properly handled and tracked until they are properly resolved or stable, and serious and unexpected events are reported to the ethics committee, competent authorities, applicants and pharmaceutical supervisory and administrative departments in a timely manner as required;
3. Major investigators regularly conduct cumulative reviews of all adverse events and, if necessary, hold researcher meetings to assess the risks and benefits of the study;

Data Preservation:

The experimental data is stored in Access database and stored locally after entering electronic data. This clinical trial uses the subject's Research Medical Record as the original data source. Researchers need to record the subject's data in the Case Report Form according to the Research Medical Record. The sponsors will verify the integrity, accuracy and authenticity of the data in Case Report Form.After completing the enrollment, complete Case Report Form is required and the first Case Report Form copy is withdrawn by the sponsor.At the end of the study, the original data, informed consent and remaining Case Report Form data will be kept at the various research centers as required.The retention period was 10 years after the end of the clinical trial.

Statistical analysis was performed by double-sided test, with P < 0.05 being statistically significant except for those specified in particular; measurements were described by means, medians, standard deviations, maximum and minimum values; counts or ranks were expressed by frequency and frequency.

Statistical Processing:

Homogeneity between groups was compared by t test, chi-square test or rank sum test.

Efficacy evaluation: Continuous corrected chi-2 test was used to compare the intracranial infection rates within 365 days after surgery. The unilateral 95% confidence interval of difference between the two groups was calculated. If the lower limit of the confidence interval was greater than -10%, the superiority was established, that is, the experimental group was superior to the control group.

Sample Size and Research Plan:

Statistical analysis uses Statistical Product and Service Solutions(SPSS) 26.0 software, the analysis process is all programmed.

The trial was designed for superiority and inferiority according to "Chow, S.C., Shao, J., and Wang, H. 2008. Sample Size Calculations in Clinical Research, Second Edition. Chapman & Hall/CRC. Boca Raton,Florida. "The main efficacy indicators were the intracranial infection rate in one year after operation. The estimated infection rate was 2.8% in the experimental group and 9.5% [18] in the control group. The other relevant parameters were set as follows: Class I error alpha=0.05 (unilateral), test efficiency 1-beta=0.8, and the number of cases in the experimental group and the control group was designed as 1:1.Comparing sample size calculation formulas based on two sample rates:

To calculate the sample size, 156 cases in the experimental group and 156 cases in the control group were obtained. Considering the dropout rate of no more than 15%, 180 cases in the experimental group and 180 cases in the control group were planned to be enrolled. The total number of cases in the two groups was 360.This study requires at least 360 patients to have sufficient test intensity to avoid false negative. In the design of the study, 600 patients were initially recruited, of whom 200 were from our center and 400 were from other centers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, regardless of gender.
2. Patients with hydrocephalus of high, normal and low pressure caused by various reasons need V-P shunt and meet the operation indications.
3. Before the start of the trial, a written informed consent signed by the subject himself or his legal representative must be obtained.

Exclusion Criteria:

1. Patients who had participated in clinical trials of other drugs or medical devices within 6 months.
2. Patients with abnormal coagulation mechanisms or who had received treatment with thrombolytic agents, anticoagulants, or inhibitors of platelet coagulation within 2 weeks, and patients with hemophilia.
3. Patients with severe diseases of other systems, such as severe diseases of the hematological, respiratory, digestive, and urinary systems, were combined.
4. Patients with co-existing infectious diseases.
5. Pregnant, lactating female patient.
6. Physicians judged other situations in which they could not participate in the trial.
7. The subjects themselves or their legal surrogates refused to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperation Intracranial infection | 10 days post-operation to 12 month post-operation
  post-operation intracranial infection(diagnosed by lumbar puncture)
Rate of postoperation Intra-abdominal infection | 10 days post-operation to 12 month post-operation
  Post-operation abdominal-cavity infection(diagnosed by WBC counting and clinical feature)

SECONDARY OUTCOMES:
Rate of Ventriculoperitoneal shunt malfunction | 10 days post-operation to 12 month post-operation
  jammed or over draining of the shunt
Rate of postoperation Surgical wound infection | 10 days post-operation to 12 month post-operation
  infection of surgical site, while intracranial and intraabdominal infection can be excluded.

OTHER OUTCOMES:
Barthel Index of activities of daily living | prior operation and 6\12 month time point
  assess patients capability of activities of daily living
Glasgow coma scale(GCS) | prior operation and 10 days post-operation to 12 month post-operation
  assess post-traumatic hydrocephalus patient's conscious status

CONTACTS AND LOCATIONS:
Overall Officials: Baiyun Liu, Ph.D, Study Chair — Beijing Tiantan Hospital affiliate to Capital Medical University
Locations (1):
- Beijing TianTan Hospital affliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Y, Green NL, Wrensch MR, Zhao S, Gupta N. Ventriculoperitoneal shunt complications in California: 1990 to 2000. Neurosurgery. 2007 Sep;61(3):557-62; discussion 562-3. doi: 10.1227/01.NEU.0000290903.07943.AF. PMID 17881969
- [Background] McGirt MJ, Zaas A, Fuchs HE, George TM, Kaye K, Sexton DJ. Risk factors for pediatric ventriculoperitoneal shunt infection and predictors of infectious pathogens. Clin Infect Dis. 2003 Apr 1;36(7):858-62. doi: 10.1086/368191. Epub 2003 Mar 18. PMID 12652386
- [Background] Choux M, Genitori L, Lang D, Lena G. Shunt implantation: reducing the incidence of shunt infection. J Neurosurg. 1992 Dec;77(6):875-80. doi: 10.3171/jns.1992.77.6.0875. PMID 1432129
- [Background] Rozzelle CJ, Leonardo J, Li V. Antimicrobial suture wound closure for cerebrospinal fluid shunt surgery: a prospective, double-blinded, randomized controlled trial. J Neurosurg Pediatr. 2008 Aug;2(2):111-7. doi: 10.3171/PED/2008/2/8/111. PMID 18671615
- [Background] Working Group on Neurosurgical Outcomes Monitoring; Woo PY, Wong HT, Pu JK, Wong WK, Wong LY, Lee MW, Yam KY, Lui WM, Poon WS. Primary ventriculoperitoneal shunting outcomes: a multicentre clinical audit for shunt infection and its risk factors. Hong Kong Med J. 2016 Oct;22(5):410-9. doi: 10.12809/hkmj154735. Epub 2016 Aug 26. PMID 27562986
- [Background] Erps A, Roth J, Constantini S, Lerner-Geva L, Grisaru-Soen G. Risk factors and epidemiology of pediatric ventriculoperitoneal shunt infection. Pediatr Int. 2018 Dec;60(12):1056-1061. doi: 10.1111/ped.13709. Epub 2018 Dec 10. PMID 30290047
- [Background] Yang YN, Zhang J, Gu Z, Song YL. The risk of intracranial infection in adults with hydrocephalus after ventriculoperitoneal shunt surgery: A retrospective study. Int Wound J. 2020 Jun;17(3):722-728. doi: 10.1111/iwj.13331. Epub 2020 Feb 19. PMID 32073232